CLINICAL TRIAL: NCT01387776
Title: Study for the Evaluation of the Benefits of 1 st Trimester Risk Markers in Detecting Early Onset Pre-eclampsia and the Use of the Placental Growth Factor (PlGF) as a Potential Marker for Trisomy 21 and Other Aneuploidies
Brief Title: Detecting Early Onset Pre-eclampsia and Use of Placental Growth Factor (PlGF) for Marker of Trisomy 21
Acronym: PlGF
Status: Terminated | Type: Observational
Why Stopped: The technique has been approved and validated
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: B-PRN-10-01
Record Dates: First submitted 2011-01-31; First posted 2011-07-06 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- study group: patients coming to clinique OVO in the 1st trimester of pregnancy to undergo prenatal screening

SUMMARY:
This is a study for the evaluation of the benefits of 1 st Trimester risk markers in detecting Early Onset Pre-eclampsia and the use of the Placental Growth factor(PIGF) as a potential marker for Trisomy 21 and other aneuploidies.

Aim of this prospective nonprofit study is to analyze the benefits of early onset pre eclampsia risk assessment in the 1st trimester (measuring biochemical markers [PIGF], blood pressure and Doppler ultrasound), and how the results can permit to modify or influence the course of the preeclampsia during the pregnancy. The investigators will also evaluate the potential use of the PIGF as a marker to improve the prenatal screening with the currently used nuchal translucency, serum Pregnancy-associated plasma protein A (PAPP-A) and free beta subunit of human chorionic gonadotropin (fBhCG) parameters.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Nulliparous pregnancy
* Gestation age between 6.0-13.6 weeks by last menstrual period verified by ultrasound
* Blood sample provided at gestational age 6.0-13.6 weeks
* Informed Consent

Exclusion Criteria:

* Multi-fetal pregnancy
* Primiparous or multiparous pregnancy
* Mental retardation or other mental disorders that impose doubts regarding the true patient's willingness to participate in the study
* Gestation age below 6.0 or above 13.6 weeks by last menstrual period verified by ultrasound.
* Lack of blood sample at the specified enrollment period
* Known major fetal anomaly or fetal demise
* Lack of demographic data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women in 1st trimester of pregnancy coming to clinique OVO for prenatal screening
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
levels of Placental Protein 13 (PP13) , PIGF, PAPP-A, PIBF | 6-13.6 wks gestation
  levels of PP13, PIGF, PAPP-A will de considered in association with Doppler ultrasound and standardised blood pressure measurements to see if they can be used as early risk markers in patients having a delivery before 34 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hemmings, MD, Principal Investigator — Clinique Ovo; Bernard Couturier, MD, Study Director — Clinique Ovo; Dominique Berube, PhD, Study Chair — Clinique Ovo
Locations (1):
- OVO Prénatal, Montreal, Quebec, Canada